CLINICAL TRIAL: NCT05812118
Title: A Classroom-based Randomized Controlled Trial to Promote Physical Literacy in Children: ALPHYL Study Protocol
Brief Title: A Classroom-based Intervention to Promote Physical Literacy in Children: ALPHYL Study Protocol
Acronym: ALPHYL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UV1564606
Record Dates: First submitted 2023-03-14; First posted 2023-04-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-03

CONDITIONS: Physical Activity
Keywords: Physical Literacy; Academic Achievement; Cognitive Function; Children; School-based Intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A classroom-based randomised controlled trial
Who Masked: Participant
Masking Description: Participants will not be aware of whether or not they received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group
- Experimental group (Experimental): Physical active learning intervention
  Interventions: Behavioral: Physical active learning

INTERVENTIONS:
Behavioral: Physical active learning — The intervention will last for 8-10 weeks. The ALPHYL intervention will be conducted in physical education (PE) and non-PE lessons by teachers. In addition to the PE lessons, at least three physically active activities in subjects other than PE will be conducted every day (5 days per week), with a total duration of approximately 30 minutes of light and moderate-to-vigorous physical activity per day. The weekly dose of physically active learning will thus be 100-150 minutes, so that a volume of 800-1200 minutes is foreseen during the 8-10 weeks. The PE classes will also be conducted in a mix of cooperative learning, non-linear pedagogy and health-based PE.
  Arms: Experimental group

SUMMARY:
The goal of this study, named the Active Learning for PHYsical Literacy (ALPHYL) study, was to describe a multicomponent class-based physically-active learning randomized control trial (RCT) in primary school children. The main purpose was to promote children's physical literacy, academic achievement and cognitive function. The ALPHYL study is mainly based on physical literacy, active school models and Supportive, Active, Autonomous, Fair and Enjoyable principles.

DETAILED DESCRIPTION:
The ALPHYL is an 8-10-week RCT that will be conducted in six primary schools (12 classes) in Valencia and its metropolitan area. Schools will be randomly assigned to the intervention or a waiting-list control group. After a 30 h in-person training course for teachers and weekly meetings in the three months of resource preparation, the ALPHYL intervention will be conducted in physical education (PE) and non-PE lessons by teachers. The intervention consists of at least three physically active learning sessions per day plus model-based PE classes. Its feasibility will be evaluated weekly according to the Reach, Effectiveness, Adoption, Implementation, and Maintenance framework. To assess its effectiveness, a pre-test, post-test and retention (8-10 weeks after the intervention) with primary outcomes (i.e. physical activity level, motor competence, perceived motor competence and physical literacy, motivation, perceived social support, academic achievement and cognitive function), secondary outcomes and covariates will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in 5th grade (i.e., 10-11 years old).
* Schools must have at least two groups of primary school 5th grade and the teachers involved in both agree to participate.
* Each class group includes at least 75% of the participants.
* Children must not have taken part in other physical activity promotion interventions in the two previous years.

Exclusion Criteria:

• None.

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change of the actual motor competence | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Assessment of the actual motor competence using Canadian Agility Movement Skill Assessment test
Change of the physical activity level | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Assessment of the physical activity by accelerometers
Change of the perceived physical literacy | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Assessment of this variable using Physical Literacy for Children Questionnaire. Minimum and maximum response values are from 1 to 4. Higher scores mean a better outcome.
Change of the perceived motor competence | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Assessment of this variable using Pictorial scale of Perceived Movement Skill Competence. Minimum and maximum response values are from 1 to 4. Higher scores mean a better outcome.
Change of the self-determined motivation for physical activity | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Adapted version for children of the Behavioural Regulation Exercise Questionnaire. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the perceived social support | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  The Physical Activity Family and Friends Support Scale. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the academic achievement | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Final grade scores at school
Change of the working memory | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Digit Span test
Change of the executive function | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Stroop test

SECONDARY OUTCOMES:
Change of the active commuting to/from school | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Survey adapted from Centers for Disease Control Kids-Walk-to-School programme by investigators of the International Physical Activity and the Environment Network. Participants will indicate the number of days travelling both to and from school by walking, bicycling or skateboarding in an average school week. Total number of active trips per week to and from school will be summed (range = 0-10 trips). Higher scores mean a better outcome.
Change of the body Mass Index | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  The assessment of height and weight will be use to calculate body mass index
Change of the cardiorespiratory fitness | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Assessment of this fitness component using Progressive Aerobic Cardiovascular Endurance Run test
Change of the physical activity participation (self-reported) | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Physical activity will be self-reported using Physical Activity Questionnaire for Children. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the alienation with school | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Health Behaviour in school-age children questionnaire. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the body image perception | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Children Body Figure Silhouette evaluation. Minimum and maximum response values are from 1 to 7. Higher scores mean overweight and obese appearance.
Change of the physical activity intention | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Future intention of physical activity scale. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the physical activity psychological need satisfaction according to the Self-Determination Theory at physical education | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Basic psychological needs satisfaction scale within physical education setting. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the perceived physical self-concept | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  The pictorial scale of Physical Self-Concept in Children. Minimum and maximum response values are from 1 to 4. Higher scores mean a better outcome.
Change of the sedentary behaviour | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Youth Leisure-Time Sedentary Behaviour Questionaire in minutes
Change of the school satisfaction | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Intrinsic Satisfaction Classroom Scale. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the social identity | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  Social Identity Questionnaire for Physical Education/Sport. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the knowledge related to physical activity and healthy lifestyles | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  This variable will be evaluated using the Self-Determination index. Minimum and maximum response values are from 1 to 5. Higher scores mean a better outcome.
Change of the math fluency calculation | Measured at baseline, immediately after the intervention and 8-10 weeks after the intervention
  The Spanish version of the Woodcock-Johnson III test

OTHER OUTCOMES:
School and home macro-scale neighborhood built environments | Measured at baseline
  Evaluation of the macro-scale neighborhood attributes using Geographic Information System-based data such as population density, land-use mix (green areas, commercial areas, recreational areas, etc.), distance to destinations (schools, parks, shops, etc.), intersection density, etc.
School and home micro-scale neighborhood built environments | Measured at baseline
  Evaluation of the micro-scale neighborhood attributes using Microscale Audit of Pedestrian Streetscapes-Global audit tool. Overall positive score ranges from 0 to 210. Higher scores mean a better outcome.
Internal physical school characteristics in relation to physical activity | Measured at baseline
  Evaluation of the physical school characteristics using International Study of Childhood Obesity, Lifestyle and the Environment School Audit Tool. Minimum and maximum values are from 0 to 37. Higher scores mean a better outcome.
Parental perceptions of the home neighborhood built environment | Measured at baseline
  Parental perceptions will be evaluated using Neighborhood Environment Walkability Scale for Youth. Minimum and maximum response values are from 1 to 4. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Estevan, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Romero-Martinez J, Menescardi C, Ortega-Benavent N, Montalt-Garcia S, Barnett LM, Garcia-Masso X, Estevan I. Effects of a classroom-based intervention to promote physical literacy in children: the randomized and controlled ALPHYL Study. J Sci Med Sport. 2025 Oct;28(10):833-839. doi: 10.1016/j.jsams.2025.05.006. Epub 2025 May 22. PMID 40450427